CLINICAL TRIAL: NCT06161298
Title: Microbe-host Interaction Relationship in Patients With Stroke-related Pneumonia
Brief Title: Microbe-host Interaction Relationship in Patients With Stroke-relatedPneumonia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: SAP20231201
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Stroke-related Pneumonia
Keywords: Stroke-related pneumonia; micropopulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All biological specimens (including throat swabs, sputum, blood) will be stored in the biological resource center of the study site after obtaining written informed consent from all subjects who volunteered to participate in the clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control group: age> 18, without lung disease
- NSAP group: patients with no stroke pneumonia
- SAP group: Those diagnosed with stroke-related pneumonia

SUMMARY:
This study intends to use a standardized cohort study to collect biological samples (including throat swabs, sputum and blood) from subjects eligible for inclusion, and use 16s DNA / metagenomic sequencing and metabolome technology to explore the microbial-host interaction relationship of SAP patients.

DETAILED DESCRIPTION:
Stroke-related pneumonia (SAP) is the most common complication of acute cerebral hemorrhage, and it is one of the main causes of disease aggravation, prolonged hospitalization and costs, and even death. The traditional antibiotic model proved ineffective, and new prevention and treatment methods were urgently sought.This study intends to use a standardized and rigorous cohort study to collect biological samples (including throat swabs, sputum and blood) of eligible subjects, and to explore the microbial-host interaction relationship in patients with SAP, which may provide new targets and new ideas for the prevention and control of SAP.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years old;
* Stroke was confirmed by imaging;
* Within 48 hours of onset, the onset time cannot be determined from the last normal observation;
* Glasgow Coma Scale (GCS) 7-14;
* SAP by clinical symptoms, laboratory examination or imaging confirmation, the modified CDC diagnostic criteria;
* The patient (or his / her legal representative) signs a written informed consent form.

Exclusion Criteria:

* Use of antibiotics within 4 weeks before stroke onset;
* The presence of other conditions that may interfere with the follow-up and outcome assessment (such as known significant prestroke disability, mRS score of 3-5, end-stage malignancy, and liver and renal failure);
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From December 2023 to December 2024, patients with new stroke at Guangdong Hospital of Traditional Chinese Medicine will be this study population. All eligible participants will be followed up for 90 days.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the microbiota in throat swabs and sputum | baseline, 3 days, 7 days, 14 days after enrollment, or at discharge
  Microbiota changes in each set of throat swabs and sputum will be examined using 16s DNA / metagenome sequencing.

SECONDARY OUTCOMES:
Utility-weighted modified Rankin scale score | 90 days after enrollment
  Utility-weighted modified Rankin scale score. Values range from 0 to 10: The higher the score, the better the result.
The European Quality of Life 5-Dimensional Questionnaire (EQ-5D-5L) | 90 days after enrollment
  The EQ-5D includes five dimensions of health: mobility, self-care, ability to perform daily activities, pain and discomfort, and anxiety and depression. EQ-5D-5L, including five severity levels (none, minor, moderate, severe, serious, and extreme). Value range 0-100: The higher the score, the worse the result.
Barthel-Index (BI) | 90 days after enrollment
  BI values range from 0-100: The higher the score, the better the result.
Changes in the blood plasma metabolites | baseline, 3 days, 7 days, 14 days after enrollment, or at discharge
  Ultra HPLC-tandem mass spectrometry will be used to test plasma metabolite expression in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwen Guo, Dr, Study Director — Guangdong Province Hospital of Tradtional Chinese Medicine

IPD SHARING:
Plan to Share IPD: No